CLINICAL TRIAL: NCT06134570
Title: ALDH1A1 as A Stem Cell Marker and Its Correlation With the Clinico-pathological Parameters in Invasive Mammary Carcinoma
Brief Title: ALDH1A1 Expression in Invasive Mammary Carcinoma
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Sohag University (Other)
Responsible Party: Principal Investigator, Nagwa Abd El-Sadek Ahmed, Lecturer at Pathology Department, Faculty of Medicine, Sohag University
Other Study IDs: Soh-Med-23-09-21PD
Record Dates: First submitted 2023-11-12; First posted 2023-11-18 (Actual); Last update posted 2023-11-18 (Actual); Status verified 2023-10

CONDITIONS: Breast Cancer
Keywords: breast cancer; CSCs; ALDH1A1
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Observational Model: Other | Time Perspective: Retrospective
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
ALDH1A1 isozyme oxidizes Retinaldehyde to retinoic acid, which regulates the expression of the genes involved in tumor-initiating stem-like cells, thereby initiating tumor growth and resistance to drugs.

Much emphasis has been focused on ALDH1A1 as a CSC marker. High expression of ALDH1A1 has been reported as a poor prognostic marker in several tumor types and is associated with poor patient outcomes .

DETAILED DESCRIPTION:
Breast cancer is one of the most common cancers among women. it is a heterogenous disease. several factors affect the prognosis of breast cancer. CSCs markers are one of the emerging prognostic biomarkers.

ALDH1A1 isozyme oxidizes Retinaldehyde to retinoic acid, which regulates the expression of the genes involved in tumor-initiating stem-like cells, thereby initiating tumor growth and resistance to drugs.

Much emphasis has been focused on ALDH1A1 as a CSC marker. High expression of ALDH1A1 has been reported as a poor prognostic marker in several tumor types and is associated with poor patient outcomes .

ELIGIBILITY:
Inclusion Criteria:

* Patients with invasive mammary carcinoma carcinoma and underwent surgery

Exclusion Criteria:

* Cases received pre-operative chemotherapy or radiotherapy.
* Cases with insufficient clinical data.

Sex: Female
Age Groups: Child, Adult, Older Adult
Study Population: sixty paraffin blocks of breast carcinoma collected from the archive of Pathology Department of Sohag Faculty of Medicine
Sampling Method: Non-Probability Sample
Enrollment: 60 (Estimated)
Dates: Start 2023-10-01 (Actual); Primary Completion 2024-06-01 (Estimated); Study Completion 2024-06-01 (Estimated)

PRIMARY OUTCOMES:
evaluate expression of ALDH1A1 in invasive mammary carcinoma | 4 month
  immunohistochemical study

CONTACTS AND LOCATIONS:
Locations (1):
- Faculty of Medicine, Sohag, Egypt